CLINICAL TRIAL: NCT01414257
Title: Rheumatrex High Dose Special Investigation (Regulatory Post Marketing Commitment Plan)
Brief Title: Methotrexate (Rheumatrex) High Dose Special Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3211003
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Arthritis; Rheumatoid; High Dose
Keywords: Rheumatrex; High Dose
MeSH Terms: conditions — Arthritis | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Methotrexate (MTX): Patients who receive the MTX Preparation at the dose higher than 8 mg/week for the treatment of Rheumatoid Arthritis.
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Methotrexate (MTX) — Methotrexate should be administered at the weekly dose of 6 mg orally once a week or twice or three times a week by subdividing the weekly dose into the relevant number of portions. When administering the subdivided doses, MTX should be administered at the interval of 12 hours on Day 1 to Day 2. When the weekly dose is subdivided into two portions, suspend the administration for the remaining 6 days. When the weekly dose is subdivided into three portions, suspend the administration on the remaining 5 days. Repeat this weekly cycle. The dose should be adjusted as appropriate depending on the age, symptom, tolerability, and response to the MTX Preparation in individual patients. The weekly dose should not be higher than 16 mg.
  Other Names: Rheumatrex

SUMMARY:
This Investigation is to be performed for the purpose of assessing the following information in the long-term post-marketing daily medical practice in the patients who receive REUMATOLEX 2 mg Capsule for the treatment of Rheumatoid Arthritis (RA) at the dose higher than 8 mg/week.

1. Condition of occurrence of ADRs
2. Factors considered to affect safety
3. Verification of efficacy

DETAILED DESCRIPTION:
Implemented as a Special Investigation by Central Registration System

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Rheumatrex in order to be enrolled in the survey
* Patients who receive the Rheumatrex at the dose higher than 8 mg/week for the treatment of Rheumatoid Arthritis

Exclusion Criteria:

* Patients who have been treated with Rheumatrex at the dose higher than 8 mg/week since the days when the high dose therapy for RA was not approved
* Patients who have been treated MTX other than Rheumatrex administered Rheumatrex

Ages: 17 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who receive the MTX Preparation at the dose higher than 8 mg/week for the treatment of Rheumatoid Arthritis.
Sampling Method: Probability Sample
Enrollment: 2860 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- University of Occupational and Environmental Health Hospital, Kitakyushu-shi, Fukuoka, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3211003&StudyName=Methotrexate%20%28Rheumatrex%29%20High%20Dose%20Special%20Investigation%20%28regulatory%20Post%20Marketing%20Commitment%20Plan%29%20

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methotrexate
Started | 2860
Completed | 2838
Not Completed | 22
Not completed — No Visit After First Day of Treatment | 12
Not completed — Protocol Violation | 10

BASELINE CHARACTERISTICS:
Population: Not in particular
Arm/Group | Methotrexate
Number analyzed (Participants) | 2838
Age, Customized [Number; unit: Participants]
  ≥15 to <65 years | 2014
  ≥65 years | 804
  Unknown | 20
Sex/Gender, Customized [Number; unit: Participants]
  Female | 2176
  Male | 659
  Unknown | 3
Steinbrocker Stage [Number; unit: Participants] — Stage was classified into four-grade based on below criteria by doctor at beginning. StageI:No radiological finding of osteolysis. StageII:1.Radiological finding of osteoporosis with or without mild fracture of subchondral bone. There may be mild cartilage destruction.
  2. Articular movement may be restricted, but no joint deformity StageIII:1.Osteoporosis and radiological finding of bone and cartilage destruction 2.Joint deformity such as subluxation, ulnar malposition or extension is present. There is no fibrous or osseous ankylosis.
  StageIV:Fibrous or osseous ankylosis is present.
  Participants
    Stage I (Initial) | 695
    Stage II (Medium) | 948
    Stage III (Progressive) | 613
    Stage IV (Terminal) | 524
    Unknown | 58
Steinbrocker Class [Number; unit: Participants] — Class was classified into four-grade based on below criteria by doctor at beginning.
  Class1:Complete ability to carry out all the usual duties without handicaps Class2:Adequate for normal activities despite handicap of discomfort or limited motion of one of the joints Class3:Limited to little or none of the duties of usual occupation or self-care Class4:Incapacitated, largely or wholly bed-ridden or confined to a wheelchair with little or no self-care
  Participants
    Class 1 | 794
    Class 2 | 1641
    Class 3 | 301
    Class 4 | 16
    Unknown | 86
Morbidity Period [Number; unit: Participants]
  <1 year | 443
  1 to ˂3 years | 512
  3 to ˂5 years | 313
  ≥5 years | 1148
  Unknown | 422
History of Methotrexate Therapy [Number; unit: Participants]
  ˂0.5 year | 737
  0.5 to ˂1 year | 254
  1 to ˂3 years | 547
  3 to ˂5 years | 300
  ≥5 years | 436
  Unknown | 554
  Not used Methotrexate Previously | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to methotrexate in a participant who received methotrexate.
Time Frame: 24 Weeks
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received methotrexate at least once.
Measure: Number; unit: Participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2838
Participants | 608

2. Primary Outcome: Disease Activity Score (DAS28)-4ESR
Description: Disease activity score based on 28-joint count and erythrocyte sedimentation rate (4 variables) (DAS28-4 [ESR]) was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count, ESR (mm/hour) and visual analogue scale (VAS) of general health assessed by participant or investigator. Higher score indicated more disease activity. The total scale range of DAS28-4 (ESR) , minimum is 0.0 and maximum can not be specified. DAS28-4 (ESR) >5.1 indicated high disease activity, ?3.2 to ?5.1 indicated moderate disease activity, <3.2 indicated low disease activity, and <2.6 indicated remission.
Time Frame: Baseline and 24 Weeks
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (ESR) at least once. Participants with observed DAS28-4(ESR) were included in table.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Methotrexate
Number analyzed (Participants) | 1526
Score
  At Baseline | 4.09 (1.235)
  At 24 Weeks | 3.21 (1.235)

3. Primary Outcome: Disease Activity Score (DAS28)-4CRP
Description: Disease activity score based on 28-joint count and C-reactive protein (4 variables) (DAS28-4 [CRP]) was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count, C-reactive protein (CRP, mg/dL) and VAS of general health. The total scale range of DAS28-4 (ESR) , minimum is 0.0 and maximum can not be specified. DAS28-4 (CRP) >4.1 indicated high disease activity, ≥2.7 to 4.1 indicated moderate disease activity, <2.7 indicated low disease activity, and <2.3 indicated remission.
Time Frame: Baseline and 24 Weeks
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (CRP) at least once. Participants with observed DAS28-4(CRP) were included in table.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Methotrexate
Number analyzed (Participants) | 1818
Score
  At Baseline | 3.55 (1.148)
  At 24 Weeks | 2.66 (1.076)

4. Primary Outcome: Change From Baseline in Disease Activity Score (DAS28)-4ESR
Description: Disease activity score based on 28-joint count and erythrocyte sedimentation rate (4 variables) (DAS28-4 [ESR]) was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count, ESR (mm/hour) and visual analogue scale (VAS) of general health assessed by participant or investigator. Mean change from baseline in the DAS28-4 (ESR) at Week 24 is calculated. The total scale range can not be specified.
Time Frame: Baseline and 24 Weeks
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (ESR) at least once. Participants with observed change in DAS28-4(ESR) were included in table.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Methotrexate
Number analyzed (Participants) | 1526
Score | -0.88 (1.156)

5. Primary Outcome: Change From Baseline in Disease Activity Score (DAS28)-4CRP
Description: Disease activity score based on 28-joint count and C-reactive protein (4 variables) (DAS28-4 [CRP]) was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count, C-reactive protein (CRP, mg/dL) and VAS of general health. Mean change from baseline in the DAS28-4 (CRP) at Week 24 is calculated. The total scale range can not be specified.
Time Frame: Baseline and 24 Weeks
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (CRP) at least once. Participants with observed change in DAS28-4 (CRP) were included in table.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Methotrexate
Number analyzed (Participants) | 1818
Score | -0.89 (1.117)

6. Secondary Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to methotrexate in a participant who received methotrexate. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to methotrexate was assessed by the investigator.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2838
Participants | 47

7. Secondary Outcome: Number of Participants With Treatment Related Pre-specified Important Serious Adverse Events
Description: Pre-specified important adverse events were 1) Interstitial pneumonia, 2) Pulmonary fibrosis, 3) Hepatic impairment, 4) Renal impairment, 5) Hematopoietic disorder, 6) Infection, and 7) Lymphoma. A treatment-related adverse event was any untoward medical occurrence attributed to methotrexate in a participant who received methotrexate. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to methotrexate was assessed by the investigator.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2838
Participants
  Interstitial Pneumonia | 7
  Pulmonary Fibrosis | 0
  Hepatic Impairment | 1
  Renal Impairment | 1
  Hematopoietic Disorder | 3
  Infection | 28
  Lymphoma | 4

8. Secondary Outcome: Clinical Efficacy Rate
Description: Clinical efficacy rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assesable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical effectiveness of methotrexate was assessed as "effective" or "ineffective" by the investigator. The assessment was based on the baseline condition of disease control and degree of alleviation from baseline in clinical symptoms and laboratory data.
Time Frame: 24 Weeks
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (clinical efficacy rate) at least once. Participants with observed effectiveness data were included in table.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2190
Percentage of Participants | 80.2 [78.5 to 81.9]

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Methotrexate
Serious Adverse Events (participants affected / at risk) | 69/2838
Other Adverse Events (participants affected / at risk) | 340/2838
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=2838)
Pneumonia (Infections and infestations) | 10
Pneumocystis jirovecii pneumonia (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 2
Pneumonia mycoplasmal (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Tuberculous pleurisy (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 1
Pyrexia (General disorders) | 2
Administration site reaction (General disorders) | 1
Platelet count decreased (Investigations) | 2
Helicobacter test positive (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Airway burns (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=2838)
Stomatitis (Gastrointestinal disorders) | 37
Hepatic function abnormal (Hepatobiliary disorders) | 217
Liver disorder (Hepatobiliary disorders) | 57
White blood cell count decreased (Investigations) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.